CLINICAL TRIAL: NCT01539642
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of the Sufentanil NanoTab PCA System/15 mcg (Zalviso™) for the Treatment of Post-Operative Pain in Patients After Open Abdominal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Talphera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IAP310
Record Dates: First submitted 2012-02-22; First posted 2012-02-27 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-09

CONDITIONS: Post-Operative Pain
Keywords: In patient, post operative pain; Adult post-operative inpatients who are expected to require parenteral opioid analgesia for at least 48 hours after open abdominal surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sufentanil NanoTab PCA System/15 mcg (Experimental)
  Interventions: Drug: Sufentanil NanoTab PCA System/15 mcg
- Placebo Sufentanil NanoTab PCA System (Placebo Comparator)
  Interventions: Drug: Placebo Sufentanil NanoTab PCA System

INTERVENTIONS:
Drug: Sufentanil NanoTab PCA System/15 mcg — 15 mcg Sufentanil NanoTab dosed sublingually every 20 minutes as needed for pain for up to 48 hours. Patient may elect to remain in study for up to 72 hours.
  Other Names: sufentanil sublingual microtablet system; Zalviso™
  Arms: Sufentanil NanoTab PCA System/15 mcg
Drug: Placebo Sufentanil NanoTab PCA System — Placebo NanoTab dosed sublingually every 20 minutes as needed for pain for up to 48 hours. Patient may elect to remain in study for up to 72 hours.
  Arms: Placebo Sufentanil NanoTab PCA System

SUMMARY:
The purpose of this study is to compare the efficacy and safety of the Sufentanil NanoTab PCA System/15 mcg to the Placebo Sufentanil NanoTab PCA System for the management of acute moderate to severe post-operative pain after open abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who are 18 years or older
* Patients who are scheduled to undergo an open abdominal surgery (including laparoscopic-assisted) under general anesthesia or spinal anesthesia that does not include intrathecal opioids during the operation.
* Post-surgical patients who have been admitted to the PACU and are expected to remain hospitalized and to have acute post-operative pain requiring parenteral opioids for at least 48 hours after surgery.

Exclusion Criteria:

* Patients who have taken an opioid for more than 30 consecutive days, at a daily dose of more than 15 mg of morphine (or equivalent), within the past 3 months prior to surgery (e.g. more than 3 doses per day of Vicodin®, Norco®, Lortab® with 5 mg hydrocodone per tablet).
* Patients with an allergy or hypersensitivity to opioids.
* Female patients who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Palmer, M.D., PhD, Study Director — Talphera, Inc
Locations (12):
- United States (12):
  - Surgical Associates of Mobile, Mobile, Alabama
  - Caring Clinical Research Corporation, Laguna Hills, California
  - The Stamford Hospital, Stamford, Connecticut
  - G&G Research, Vero Beach, Florida
  - Rush Pain Center, Chicago, Illinois
  - CRC of Jackson, Jackson, Mississippi
  - Cooper University Hospital, Camden, New Jersey
  - Phoenix OB GYN Associates, Moorestown, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Duke University Medical Center, Durham, North Carolina
  - Jefferson Hospital, Philadelphia, Pennsylvania
  - Memorial Hermann -Memorial City Medical Center, Houston, Texas

REFERENCES:
- [Background] Ringold FG, Minkowitz HS, Gan TJ, Aqua KA, Chiang YK, Evashenk MA, Palmer PP. Sufentanil sublingual tablet system for the management of postoperative pain following open abdominal surgery: a randomized, placebo-controlled study. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):22-30. doi: 10.1097/AAP.0000000000000152. PMID 25318408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period of 10 months - March 1, 2012 to December 28, 2012; Recruitment and screening occurred at clinical research centers and hospitals.
Pre-assignment Details: Patients were excluded per protocol exclusion criteria at Screening as well as post surgery for certain issues including the following:
  1. Patients who were not awake or stable
  2. Patients with arterial oxygen saturation that couldn't be maintained at 95% or greater
  3. Patients with uncontrollable vomiting
Groups:
- Sufentanil NanoTab PCA System/15 mcg: Sufentanil NanoTab PCA System/15 mcg : 15 mcg Sufentanil NanoTab dosed sublingually q 20 minutes as needed for pain for at least 48 hours and up to 72 hours
- Placebo Sufentanil NanoTab PCA System: Placebo Sufentanil NanoTab PCA System : Placebo NanoTab dosed sublingually q 20 minutes as needed for pain for at least 48 hours and up to 72 hours
Period: Overall Study
Arm/Group | Sufentanil NanoTab PCA System/15 mcg | Placebo Sufentanil NanoTab PCA System
Started | 114 | 58
Completed | 78 | 27
Not Completed | 36 | 31
Not completed — Lack of Efficacy | 20 | 18
Not completed — Patient ready for early discharge | 8 | 7
Not completed — Adverse Event | 6 | 4
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Sufentanil NanoTab PCA System/15 mcg: Sufentanil NanoTab PCA System/15 mcg : 15 mcg Sufentanil NanoTab dosed sublingually q 20 minutes as needed for pain for at least 48 hours. Patient may elect to remain in study for up to 72 hours
- Placebo Sufentanil NanoTab PCA System: Placebo Sufentanil NanoTab PCA System : Placebo NanoTab dosed sublingually q 20 minutes as needed for pain for at least 48 hours. Patient may elect to remain in study for up to 72 hours
- Total: Total of all reporting groups
Arm/Group | Sufentanil NanoTab PCA System/15 mcg | Placebo Sufentanil NanoTab PCA System | Total
Number analyzed (Participants) | 114 | 58 | 172
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 91 | 36 | 127
  >=65 years | 23 | 22 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (13.5) | 57.4 (14.9) | 55.2 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 49 | 128
  Male | 35 | 9 | 44
Region of Enrollment [Number; unit: participants]
  United States | 114 | 58 | 172

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Summed Pain Intensity Difference (SPID) Over the 48-hour Study Period (SPID-48).
Description: SPID-48 is the sum of the pain intensity difference (PID) over the 48 hour time period. A pain intensity score of 0 (no pain) to 10 (worse possible pain) is obtained before starting the study and throughout the 48 time period. The pain score at each assessment time is subtracted from the baseline pain score to provide the total sum score or SPID-48. A higher SPID-48 is better and indicates a reduction in pain intensity compared to the baseline score. The range of SPID48 scores were -232 to 326.
  Time-weighted SPID48 = ∑ [T(i) - T(i-1)] x PID(i), where T(0) = Time 0 (baseline), T(i) is the scheduled or unscheduled assessment time, and PID(i) is the PID score at time i for i=0 to 48 hours.
  Note: Active group n=114 and placebo group n=58, instead of active n=115 and placebo n=57, due to one "active" patient receiving placebo inadvertently.
Time Frame: 48 hours
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Sufentanil NanoTab PCA System/15 mcg | Placebo Sufentanil NanoTab PCA System
Number analyzed (Participants) | 114 | 58
Units on a scale | 105.60 (10.14) | 55.58 (13.11)
Statistical Analysis 1: Comparison: Sufentanil NanoTab PCA System/15 mcg vs Placebo Sufentanil NanoTab PCA System; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = 50.02, 95% CI 2-sided [19.89 to 80.14], Standard Error of Mean 15.25

ADVERSE EVENTS:
Time Frame: Treatment period of 48 hours (patients could elect to stay in study up to 72 hours). AEs collected from time of first dose of study drug through 12 hours after last dose of study drug.
Arm/Group | Sufentanil NanoTab PCA System/15 mcg | Placebo Sufentanil NanoTab PCA System
Serious Adverse Events (participants affected / at risk) | 1/114 | 0/58
Other Adverse Events (participants affected / at risk) | 26/114 | 15/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sufentanil NanoTab PCA System/15 mcg (N=114) | Placebo Sufentanil NanoTab PCA System (N=58)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — Investigator deemed event was unrelated to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sufentanil NanoTab PCA System/15 mcg (N=114) | Placebo Sufentanil NanoTab PCA System (N=58)
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0
Chest Pain (General disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 1
Hypertension (Vascular disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 16 | 13
Oxygen Saturation Decreased (Investigations) | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0
Tachycardia (Cardiac disorders) | 2 | 0 — All adverse events in this table were assessed by the PI as possibly or probably related to study drug
Vomiting (Gastrointestinal disorders) | 4 | 2
Pyrexia (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days